CLINICAL TRIAL: NCT00221585
Title: The National Danish Schizophrenia Project
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: University of Aarhus (Other)
Other Study IDs: 5490-184
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2006-11-07 (Estimated); Status verified 1997-07

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Behavioral: Psychosocial treatment/Psychodynamic treatment

SUMMARY:
A prospective, longitudinal, multi-centre investigation (16 centres), including 562 patients, consecutively referred during two years, with a first-episode psychosis of ICD-10, F-2 type. Patients were treated with: 1) 'Supportive psychodynamic psychotherapy as a supplement to treatment as usual', 2) an 'Integrated, assertive, psychosocial and educational treatment programme', and 3) 'Treatment as usual'.

DETAILED DESCRIPTION:
The study is a prospective, comparative, longitudinal study with an intervention period of a minimum of two years and a registration of data at baseline and 1, 2 and 5 years after inclusion. Three sub-cohorts with different treatment modalities were designed:

Treatment1: 119 patients were, in addition to TaU, offered SPP, i.e. a scheduled manualised supportive individual psychotherapy (1 session of 45 min. per week, for a period of 1-3 years) and/or group psychotherapy (1 session of 60 min. per week for a period of 1-3 years). Anti-psychotic medication was given in doses based on individual needs; Treatment 2: 139 patients were offered IT, i.e. a scheduled, two-year long programme consisting of assertive community treatment, psycho-educational multi-family treatment (a.m. McFarlane, consisting of 4-6 families including the patients, meeting 1½ hour every second week for 1½ year), social skills training (concerning medication, self-management, coping with symptoms, conversational skills, problem and conflict solving skills), and antipsychotic medication (low dose strategy). This project, OPUS, has been described in detail elsewhere

ELIGIBILITY:
Inclusion Criteria:

consecutively referred patients, age 16-35 years, who suffered from a first-episode psychosis of the schizophrenic spectrum disorder (ICD-10, DF 20-29).

-

Exclusion Criteria:

* patients suffering from mental retardation or other organic brain damage, and patients who were not proficient enough in Danish due to their foreign origins.

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1997-10; Study Completion 2005-07

CONTACTS AND LOCATIONS:
Overall Officials: Bent Rosenbaum, DMSci, Study Director — Psychiatric Center Glostrup, Dernmark
Locations (1):
- Psychiatric Hospitäl in Aarhus, Risskov, Aarhus, Denmark

REFERENCES:
- [Result] Rosenbaum B, Valbak K, Harder S, Knudsen P, Koster A, Lajer M, Lindhardt A, Winther G, Petersen L, Jorgensen P, Nordentoft M, Andreasen AH. The Danish National Schizophrenia Project: prospective, comparative longitudinal treatment study of first-episode psychosis. Br J Psychiatry. 2005 May;186:394-9. doi: 10.1192/bjp.186.5.394. PMID 15863743